CLINICAL TRIAL: NCT03585283
Title: Effects of Myofascial Releasing on Neck Pain in Patients With Trigger Points: A Single Blinded, Randomized Controlled Trial
Brief Title: Effects of Myofascial Releasing on Neck Pain in Patients With Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Ms.C Research Assistant, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AbantIBU-Phys2
Record Dates: First submitted 2018-06-20; First posted 2018-07-13 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Trigger Point Pain, Myofascial; Neck Pain
Keywords: Myofascial Release; Manual Therapies
MeSH Terms: conditions — Myofascial Pain Syndromes; Neck Pain

STUDY DESIGN:
Intervention Model Description: Patients' information and contact will be obtained from physiatrist and willing participant's gender, age and pain onset data will be processed with a random number generator in order to form groups. Patients will divide randomly into two groups as intervention and control with a normal distribution of gender, age and pain onset.
Who Masked: Participant, Outcomes Assessor
Masking Description: Intervention group will receive myofascial release and control group will receive a sham therapy by using same treatment and handling position without applying myofascial release techniques.
  Participant will be evaluated at baseline, 4 weeks later and 12 week later by an another investigator who does not aware of groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Group (Experimental): Myofascial release will be applied by physiotherapist two times a week for four weeks which is a manual therapy technique includes stretching and compression of soft tissues according to fascial chains.Each session will be approximately 45 min long. Participant will be reevaluated 8 week later after last session for a follow-up assessment.
  Interventions: Other: Myofascial Group
- Sham Group (Sham Comparator): Sham application will be applied two times a week for four weeks. Each session will be approximately 45 min long. Participant will be reevaluated 8 week later after last session for a follow-up assessment.
  Interventions: Other: Sham Group

INTERVENTIONS:
Other: Myofascial Group — Manual myofascial release will be applied at prone position. Patient's upper thoracic and cervical region will be undressed. Researcher will use direct and indirect myofascial release techniques on upper thoracic and cervical region focusing on trigger point located muscles (most frequently m. trapezius)
  Arms: Myofascial Group
Other: Sham Group — Patient's upper thoracic and cervical region will be undressed. Researcher will place his hands on points that used for myofascial release however no pressure or release techniques will be used.
  Arms: Sham Group

SUMMARY:
Aim of this study is to investigate effectiveness of myofascial releasing on neck pain related to trigger points located on upper cervical region.

DETAILED DESCRIPTION:
Neck pain is the second most common musculoskeletal pain after lumbar pain. Prevalence is 27.2% female and 17.4% in male population. Approximately 1/3 of acute onset neck aches become chronic. It causes increasing the cost of treatment and also the loss of labor.

Myofascial pain is usually considered caused by myofascial trigger points. The trigger points in the neck muscles have been associated with a possible source of referred facial and cranial pain. Mechanical neck pain is a non-radicular pain caused by local musculoskeletal structures and is characterized by a spasm of the cervical muscles. Posture, emotional stress, cold and fatigue are etiologic causes, and pain is also reflected to the cervical, occipital and scapular regions depending on the severity of muscle spasm and the presence of trigger point in myofascial pain syndrome.

Myofascial releasing is a specific type of passive soft tissue mobilization. Triggers points often considered as a pathology that occurs after excessive load or trauma on soft tissue which disturbs blood circulation. Fascial restriction can be found with triggers points and taut band.

In this study effects of myofascial release on triggers points will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Non specific cervical pain
* Symptoms should last longer than 4 weeks
* Palpable trigger points on upper thoracic region

Exclusion Criteria:

* Cervical radiculopathy
* Previous manual therapy treatment history
* Sensory or motor function loss
* Rheumatologic diseases
* Structural damage on cervical spina
* Trauma history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-08-12 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Assessment of Pain Pressure Threshold on Trigger Points with Algometer | 12 weeks
  Trigger points will be located with palpation and with slight pressure most painful one will be marked. Pressure will be applied by researcher and patient will be informed to notify researcher immediately after starting to feel pain from pressure.

SECONDARY OUTCOMES:
Neck Disability Index | 12 weeks
  The Neck Disability Index will be used to record perceived disability according to patients with neck pain. Neck disability index is a 10 question self administrated questionaire. Each question scored from 0-5 for a total of 50 point.
Assessment of Perceived Pain on Cervical Region | 12 weeks
  Visual analog scale (VAS) will be used to assess patients' pain while doing neck rotations. Patients will mark their perceived pain on a 10 cm horizontal line. Left side of line considered as 0 (no pain at all) and right side considered as 10 (most intense pain experienced so far).
Global Rating of Change Scale-Turkish Version | 12 weeks
  Patients global perception on effects of treatment will be assessed with a 9 aspect scale. 5 was considered as no change from the baseline and 1-4 indicate decline in symptoms and 6-9 indicate improvement.
Assessment of Cervical Active Range of Motion (ROM) | 12 weeks
  Patients cervical flexion, lateral flexin and rotation ROM's will be assessed with a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Şebnem Avcı, Ph.D, Study Director — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No